CLINICAL TRIAL: NCT02874677
Title: Effects of an Endurance Training Program at Ventilatory Threshold on the Walking Distance of Ambulatory Patients With Multiple Sclerosis
Brief Title: A Reeducation Program to Effort to Improve the Walking of Multiple Sclerosis Patients
Acronym: AEROSEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: material issues in study centres
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC-P0048; 2016-A00745-46 (Other: ANSM)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Ventilatory threshold; Effort Reeducation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Routine activities
- Experimental (Experimental): Effort reeducation program : 3 sessions of 20 minutes per week during 6 weeks
  Interventions: Other: Effort reeducation program

INTERVENTIONS:
Other: Effort reeducation program — personalized reeducation program at a load level preceding hyperventilation
  Arms: Experimental

SUMMARY:
Multiple sclerosis (MS) is a disease affecting the white matter of the central nervous system. In France, it concerns approximately 80 000 patients and represents one of the most frequent neurological affections in young adults. Effort deconditioning of people affected by MS is already proven, but it is not just linked to the disease itself. The decrease of capacities to produce an effort is aggravated by neurovegetative and cardiovascular disorders. The limitation or the complete stop of physical activity is often linked to the fear of a handicap aggravation. Causes of stop are multiple, including fatigue and balance disorders, even if the handicap level is low (average EDSS = 2). Walking disorders generated by MS are frequent, represent the first symptom of the disease (10 to 20 % of cases) and alter significantly the quality of life.

Some reeducation programs were proposed in hospitalization with some efficiency on functional capacities. It is now admitted that physical exercise is not noxious, and allows the implementation of effort reeducation for MS. Randomized controlled studies have shown in MS patients an improvement of physical abilities, of O2max (aerobic capacity), of quality of life and a decrease of fatigue. For MS, only a few studies estimate the effect of effort reeducation on treadmill. Unfortunately, the efficiency of these programs on walking endurance are controversial.

During the maximal cardiorespiratory effort test, the ventilatory threshold 1 (VT1) corresponds to a greater increasing of CO2 compared to O2. The identification of VT1 allows the precise determination of the limit from which the body is incapable of producing the necessary energy to realize an effort using the aerobic metabolism. The VT1 is situated at a level of load with enough intensity for the subject to support the test without dyspnea. A VT1 lower than 40 % of the theoretical VO2 max is considered as a marker of maladjustment to effort due to dyspnea and excessive muscular fatigue. This indication is very informative about the quality of life of patients.

The goal of this study is to apply a personalized reeducation concerning the working load pre-hyperventilation to deconditioned subjects, easily worried by effort induced breathlessness and fatigue in order to get the optimization of the aerobic function. The hypothesis is that reeducation at this level improves the distance of walking and the quality of life of patients affected by MS.

DETAILED DESCRIPTION:
Multiple sclerosis is a disease affecting the white matter of the central nervous system. In France, it concerns approximately 80 000 patients and represents one of the most frequent neurological affections in young adults. There are several symptoms, including pyramidal syndrome, sensory syndrome, visual disorders, fatigue, bladder-sphincter disorders, etc. It is an unpredictable chronic disease. Most of the time, it evolves by relapse at the beginning, then, after a few years, the disease becomes secondarily progressive. In some cases, the evolution is directly progressive.

Efforts oriented to the deconditioning of people affected by multiple sclerosis are already proven, but they are not only linked to the disease itself. The decrease of capacities to produce an effort is aggravated by neurovegetative and cardiovascular disorders.

The limitation, even the complete stop, of physical activity is often linked to the fear of a handicap aggravation. Causes of stop are multiple, including fatigue (general and muscular) and balance disorders, even if the handicap level is low (average EDSS = 2).

Walking disorders generated by this pathology are frequent and represent the first symptom of the disease (10 to 20 % of cases). These walking disorders quickly appear and alter significantly the quality of life.

After several years of evolution, functional effects are more and more pronounced. The walking perimeter is estimated at 500 meters without help after 7 years of evolution on average, and no more than 100 meters after 15 years of evolution. At this stage, 50 % of patients need a technical help to move.

Some reeducation programs were proposed in hospitalization with some efficiency on functional capacities. It is now admitted that physical exercise is not noxious, and allows the implementation of effort reeducation for this pathology. Randomized controlled studies have shown in multiple sclerosis patients an improvement of physical abilities, of O2max (aerobic capacity), a decrease of fatigue and an improvement of quality of life.

Actually, the cyclo-ergometer is the most common device used for the effort reeducation. Another approach is the use of a treadmill, based on the improvement of the walking reflex modeling and the enhancement of the specific walking work, thanks to a high frequency of repetitions. This device seems more adapted for the improvement of walking disorders than the cyclo-ergometer.

For this pathology, only a few studies estimated the effect of effort reeducation on treadmill. Unfortunately, the efficiency of these programs on walking endurance is not well known and results are controversial. Indeed, only two randomized, controlled trials showed improvements of the walking speed and the energy cost of walking.

However, the impact on the 2-Minute Walk Test (2MWT) was contradictory, probably due to the population studied (different EDSS and age) and the training duration (4 weeks Vs 8 weeks). Moreover, in these studies, the effort intensity is most of time determined from an arbitrary percentage of the theoretical maximal heart rate (HR) or the VO2max.

The heart rate corresponding to the level of load of the ventilatory threshold (VT) described by Wasserman and al (1973) could be more efficient to measure the intensity of reeducation, compared to a heart rate (HR) determined from an arbitrary percentage. Four reasons are highlighted:

1. The ventilatory threshold represents a well defined metabolic level (individualized measure)
2. According to the subjects, ventilator threshold is not a constant percentage of "O2max", and suggests that it is also an individualized measure.
3. During the maximal cardiorespiratory effort test, the ventilatory threshold 1 (VT1) corresponds to a greater increasing of CO2 compared to O2. The identification of this threshold allows the precise determination of the limit from which the body is incapable of producing the necessary energy to realize an effort using the aerobic metabolism.
4. The VT1 is situated at a level of load with enough intensity for the subject to support the test without dyspnea. A VT1 lower than 40 % of the theoretical VO2 max is considered as a marker of maladjustment to effort due to dyspnea and excessive muscular fatigue. This indication is very informative about the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* People with remittent or progressive multiple sclerosis defined by the criteria of Mc Donald revised in 2005
* Expended Disability Status Scale (EDSS) between 4 and 6
* Age between 18 and 65 years old
* No defined relapse of MS for at least 6 weeks
* At least more than 4 weeks since the last corticoids bolus
* Coverage of the social insurance

Exclusion Criteria:

* Understanding disorders
* Medical history of orthopaedic or and rheumatologic invalidating
* Contraindications to test effort, after a cardiological consultation and ECG
* Cardiovascular and respiratory diseases not stabilized
* Osteo-articular diseases not stabilized
* Pregnant or breast-feeding woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Distance estimated by the 6 minutes Walk Test | Change in baseline at 6 weeks and at 3 months
  Distance covered during 6 minutes estimated by the 6 minutes Walk Test (6MWT) performed at the inclusion visit then at 6 weeks and at 3 months after the effort reeducation program (experimental group) or not (control group).

SECONDARY OUTCOMES:
Walking speed measured by the timed 25-ft walk test (T25FWT) | Change in baseline at 6 weeks and at 3 months
Heart rate estimation at the end of the 6 minutes walk test | Change in baseline at 6 weeks and at 3 months
Walking perception measured by the Twelve Item MS Walking Scale (MSWS-12) scale | Change in baseline at 6 weeks and at 3 months
  It is an auto-questionnaire which estimates the impact of the disease on the walk capacity.
Effort test for the estimation of the maximal consumption of oxygen (O2max) | Change in baseline at 6 weeks and at 3 months
Multiple sclerosis-59 French scale for the estimation of the quality of life | Change in baseline at 6 weeks and at 3 months
Fatigue Impact Scale (EMIF-SEP) | Change in baseline at 6 weeks and at 3 months
Effort test for the estimation of the ventilatory threshold (VT1) | Change in baseline at 6 weeks and at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Massot, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (4):
- France (4):
  - Centre Hospitalier Universitaire d'Amiens, Amiens, Hauts-de-France
  - Centre Jacques Calvé, Berck, Hauts-de-France
  - Centre Hospitalier Régional Universitaire de Lille, Lille, Hauts-de-France
  - Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille, Hauts-de-France

IPD SHARING:
Plan to Share IPD: No